CLINICAL TRIAL: NCT01116440
Title: A Double Blind, Randomized, Controlled, Multicenter, Efficacy and Safety Study of Oral BGS649 vs. Placebo (Each Co-administered With a Combined Oral Contraceptive) Assessing Pain Response in Patients With Refractory Endometriosis
Brief Title: A Safety & Efficacy Study of BGS649 in Women With Refractory Endometriosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBGS649A2202
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Pelvic Pain Associated With Refractory Endometriosis
Keywords: Menstrual pain; Refractory endometriosis; Pelvic pain
MeSH Terms: conditions — Dysmenorrhea; Endometriosis; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BGS649 co-administered with Levora 28™ (Experimental)
  Interventions: Drug: BGS649
- Placebo co-administered with Levora 28™ (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGS649 — 0.1 mg capsules for oral administration. A total dose of 3 capsules of BGS649 0.1mg will be administered at randomization, week 4, and week 8 at the study site.
  Arms: BGS649 co-administered with Levora 28™
Drug: Placebo — Placebo matching BGS649 will be provided by Novartis as capsules for oral administration. Three capsules of placebo will be administered at randomization, week 4, and week 8 at the study site.
  Arms: Placebo co-administered with Levora 28™

SUMMARY:
The purpose of this study is to determine efficacy, safety, tolerability and pharmacokinetics of multiple doses of BGS649 with concurrent daily administration of combined oral contraception in patients with refractory endometriosis

ELIGIBILITY:
Inclusion Criteria:

* Must have surgical diagnosis of endometriosis est. w/in 5 years before screening. Subjects must have self reported moderate to severe pelvic pain at screening to be confirmed during the run-in-phase
* Subjects with moderate to severe pelvic pain who were refractory to surgery (persistent or recurrent pelvic pain within 24 months after any therapeutic surgery) and at least two hormonal therapies from two different classes, including one approved hormonal therapy

Exclusion Criteria:

* Subjects who have undergone hysterectomy or bilateral oophorectomy.
* Surgical treatment of endometriosis within 3 months before screening.
* Subjects who are pregnant or who were pregnant within 3 months of visit one.
* Subjects who are nursing or lactating
* Subjects who are tobacco smokers.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-04-15 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2012-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkin, PhD FRCP, Study Director — Mereo BioPharma
Locations (44):
- United States (42):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Precision Trials, Phoenix, Arizona
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Center for Fertility and Women's Health, New Britain, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Zasa Clinical Research, Boynton Beach, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - University of Miami School of Medicine & Clinics, Miami, Florida
  - West Broward OB/GYN Associates, Plantation, Florida
  - Comprehensive Clinical Trials,LLC, West Palm Beach, Florida
  - Associated Pharmaceutical Research, Decatur, Georgia
  - Legacy Obstetrics & Gynecology, Decatur, Georgia
  - Minority Clinical Research Center of Atlanta, Riverdale, Georgia
  - Christie Clinic, Champaign, Illinois
  - Women's Health Practice Center, Champaign, Illinois
  - The Advanced Gynecologic Surgery Institute, Naperville, Illinois
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Green Clinic, LLC, Ruston, Louisiana
  - NECCR, Fall River, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Montana Medical Research, Missoula, Montana
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Women's Health Research Center, Plainsboro, New Jersey
  - Southwest Clinical Research, Albuquerque, New Mexico
  - New Hanover Medical Research, Wilmington, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - HWC Women's Research Center, Englewood, Ohio
  - Promedica Health System, Toledo, Ohio
  - Ilumina Clinical Associates, Hopwood, Pennsylvania
  - Medical Research South, Charleston, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Magnolia OB/GYN Research Center, Myrtle Beach, South Carolina
  - Practice Research Organization, Dallas, Texas
  - Centex Research, Houston, Texas
  - Bexar Clinical Trials, Irving, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Eastern Va Medical School, Norfolk, Virginia
  - VCU Health Systems, MCV, Richmond, Virginia
  - Valley Women's Clinic, Renton, Washington
- Puerto Rico (2):
  - Henry Rodriguez-Ginorio, MD, San Juan, Pr
  - Ponce School of Medicine, Ponce

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Started | 11 | 16
Completed | 8 | 9
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Withdrawal
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Started | 8 | 9
Completed | 8 | 7
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Follow-up
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Started | 8 | 7
Completed | 8 | 5
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set.
Groups:
- BGS649 Co-administered With Levora 28™: BGS649: 0.1 mg capsules for oral administration. A total dose of 3 capsules of BGS649 0.1mg administered at randomization, week 4, and week 8 at the study site.
- Placebo Co-administered With Levora 28™: Placebo: Placebo matching BGS649 provided by Novartis as capsules for oral administration. Three capsules of placebo administered at randomization, week 4, and week 8 at the study site.
- Total: Total of all reporting groups
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™ | Total
Number analyzed (Participants) | 11 | 16 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 16 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (5.75) | 29.4 (5.67) | 29.4 (5.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 12 | 17
  Black | 1 | 3 | 4
  Other | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 16 | 27
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (4.98) | 25.6 (4.11) | 26.6 (4.54)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Baseline to Week 12 in Numeric Rating Scale Pelvic Pain Score
Description: Mean change from baseline to Month 3 (Week 12) in Number Rating Scale pelvic pain score. The Numeric Rating Scale is a scale between 0 and 10 where 0 is no pain and 10 is the worse pain you can imagine.
Time Frame: 12 weeks
Population: Full analysis set. All patients randomised excluding those who were randomised inadvertently and did not receive study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Number analyzed (Participants) | 11 | 16
units on a scale | -0.7637 (2.12386) | -2.1706 (2.27246)

2. Secondary Outcome: Mean Change From Baseline to 4 Weeks in Numeric Rating Scale Pelvic Pain Scores
Description: Mean change from baseline in Numeric Rating Scale pelvic pain scores to 4 weeks. The Numeric Rating Scale is a scale between 0 and 10 where 0 is no pain and 10 is the worse pain you can imagine.
Time Frame: 4 weeks
Population: Full Analysis Set. All randomized patients excluding patients randomized inadvertently who did not receive drug (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Number analyzed (Participants) | 11 | 16
score on a scale | -0.6596 (1.34546) | -0.9282 (1.05794)

3. Secondary Outcome: Percentage of Patients Achieving a Response in Numeric Rating Scale Pelvic Pain Score
Description: The proportion (expressed as a percentage) of patients achieving a response in the Numeric Rating Scale pelvic pain score where a response is defined as greater than or equal to 2-point improvement from baseline or a greater than or equal to 30% improvement in the score. The Numeric Rating Scale is a scale between 0 and 10 where 0 is no pain and 10 is the worse pain you can imagine.
Time Frame: 12 weeks
Population: Full Analysis Set. All participants randomized except patients inadvertently randomized who didn't receive study drug (ITT principles)
Measure: Number; unit: percentage of participants
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Number analyzed (Participants) | 11 | 16
percentage of participants | 9.1 | 37.5

4. Secondary Outcome: Mean Change From Baseline in Numeric Rating Scale Pelvic Pain Scores
Description: Mean change from baseline in Numeric Rating Scale pelvic pain scores to 8 weeks. Where the Numeric Rate Scale Pelvic Pain Score is a scale between 0 and 10, where 0 is no pain and is the worse pain you can imagine.
Time Frame: 8 weeks
Population: Full Analysis Set. All randomized patients excluding patients randomized inadvertently who did not receive drug (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Number analyzed (Participants) | 11 | 16
score on a scale | -1.2840 (2.18569) | -2.0601 (2.11810)

5. Secondary Outcome: Percentage of Patients Achieving a Response in Their Pelvic Pain Score Measured on the Modified Biberoglu & Behrman Scale
Description: The proportion of patients (expressed as a percentage) achieving a response to their pelvic pain score measure on the Biberoglu and Behrman pelvic pain score where a response is defined as a greater than or equal to 1-point improvement from baseline. B & B scales allow for grading pain with a score between 0 and 4 with higher number being more severe pain.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Number analyzed (Participants) | 11 | 16
percentage of participants | 0 | 31.3

ADVERSE EVENTS:
Description: After unblinding the study, it was found that 1 subject in the placebo arm was dosed with BGS649 and therefore the safety population is 15 and the BGS649 arm is 12.
Arm/Group | BGS649 Co-administered With Levora 28™ | Placebo Co-administered With Levora 28™
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/15
Other Adverse Events (participants affected / at risk) | 10/12 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 Co-administered With Levora 28™ (N=12) | Placebo Co-administered With Levora 28™ (N=15)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 Co-administered With Levora 28™ (N=12) | Placebo Co-administered With Levora 28™ (N=15)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Gastroentritis viral (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Smear cervix abdominal (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Psychiatric disorders (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Mood swings (Nervous system disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Premenstrual syndrome (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
After unblinding it was found that one of the placebo patients had been given active drug. Therefore the safety populations has 12 patients on active and 15 on placebo. The study was terminated for administrative reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs must seek written permission from the sponsor prior to publication of any trial results.